CLINICAL TRIAL: NCT06787599
Title: The Effect of Synchronous Homebased Tele-exercise on Physical Function, Daily Physical Activity and Frailty in Peritoneal Dialysis Patients: A Randomized Pilot Trial
Brief Title: The Effect of Home Based Tele-Exercise on Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA25PD-2-01
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: End Stage Renal Disease; Peritoneal Dialysis Complication
Keywords: Tele-exercise; Peritoneal; Dialysis Patients; Frailty; Physical function
MeSH Terms: conditions — Kidney Failure, Chronic; Frailty

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocate to intervention group or control group and will be examined in the same way.
Who Masked: Outcomes Assessor
Masking Description: A research project collaborator who is not informed about grouping of participants will obtain outcome measurements of the functional test. Outcome adjudicators, and data analysts will be kept blinded to the allocation. Moreover, all investigators, staff, and participants will be kept masked to outcome measurements and trial results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The participants (n = 15) in the study group will be given an online personalized exercise program at home in non-peritoneal dialysis (PD). Each session will be 40 to 45 min in duration for 3 days per week over 12 weeks, 36 sessions in total.
  Interventions: Behavioral: Home-based Tele Exercise
- Control group (No Intervention): Patients allocated to the control group (n = 15) will receive their standard nephrological care. Through the 12- week period, all control participants will be instructed to maintain the standard treatment regimen and to maintain their customary dietary and physical activity patterns.

INTERVENTIONS:
Behavioral: Home-based Tele Exercise — The participants in the study group will be given an online personalized exercise program at home in non-peritoneal dialysis (PD) days. Synchronous tele-exercise will be delivered using the free teleconference application (app) (Google Meets software). The groups of teleexercises will be private and the professional will send the link for each training session and will control the access of the participants. Each session will be 40 to 45 min in duration for 3 days per week over 12 weeks, 36 sessions in total.
  Arms: Exercise group

SUMMARY:
Brief Summary:

The objective of the trial is to assess the effect of synchronous home-based tele exercise on daily activity level, functional status and frailty level in Peritoneal Dialysis patients.

Condition or disease Intervention/treatment End Stage Renal Disease Peritoneal Dialysis Complication Behavioral: Home-based Tele Exercise

DETAILED DESCRIPTION:
Patients with renal failure undergoing peritoneal dialysis (PD) therapy typically have very low levels of physical activity (PA), and this is associated with greatly increased morbidity and mortality. Although PD prevents premature death of patients, it can lead to many complications. During the years of treatment, they suffer from various problems such as malnutrition, reduced physical performance, reduced aerobic capacity, low quality of life and inactivity, so that the activity level physical activity of these patients is significantly lower than that of healthy people.

According to studies, regular exercise is beneficial for patients at all stages of renal disease, and the current recommendations for the prevention and management of side effects in PD patients, especially in the elderly, is regular exercise because it improves physical performance and PA.

There are several barriers to participation in PA for people with chronic kidney disease (CKD), especially those who are undergoing PD treatment that prevent them from adopting a consistent exercise program. These include issues specific to PD such as the risk of peritonitis, the need for aseptic technique during bag changes, and the physical discomfort associated with carrying dialysate. Personal issues that prevent participation in PA include lack of knowledge about appropriate exercise and its benefits, and lack of energy or motivation.

To increase activity levels, clinicians and researchers have experimented with different types of interventions, including home-based exercise programs, which are a suitable option for PD patients to reduce their costs and make it easy to adhere to.

Home-based exercise has the potential to utilize higher volume and higher intensity training if activity is monitored by a coach. However, many of these programs are unsupervised and this is one of the major disadvantages of home-based exercise programs. Lack of prior knowledge about the safety and benefits of exercise programs, fear of injury, and lack of interest or motivation are barriers to exercise at home.

Tele-rehabilitation is rehabilitation services provided to patients from distant locations using information and communication technologies. Tele rehabilitation consultations may include diagnosis, assessment, education, therapy, goal setting, and monitoring. Literature reviews on telerehabilitation practices in the older people have shown that tele-rehabilitation can produce results similar to face-to-face methods.

Communication between patients and rehabilitation specialists takes place through a variety of synchronous approaches such as telephony, internet-based video conferencing, or asynchronous methods like video-based exercise. E-Health interventions utilizing some of these techniques to support prostate, colorectal, breast and leukemia cancer populations have already been trialed with good effects in terms of improved PA levels and reduced sedentary behavior. Several studies have reported the use of eHealth-based self-management interventions in CKD patients.

However, further research is needed to better understand the extent to which these techniques are acceptable, safe and potentially effective for supporting individuals undergoing PD treatment, given their unique needs and risk profile, is unknown. Our study seeks to address this gap by conducting a pilot evaluation of synchronous home-based tele exercise intervention designed for PD patient.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and over
2. At least 3 months of stable peritoneal dialysis (PD) history
3. Permission from their doctors
4. Have decision-making capacity to enable them to give informed consent to take part in the study
5. Have access to a smart device (e.g., smartphone, laptop or tablet), and have internet access

Exclusion Criteria:

1. Unstable cardiac status, including angina, decompensated congestive heart failure, or uncontrolled arrhythmias
2. Active infection or acute medical illness
3. Hemodynamic instability
4. Labile glycemic control
5. Individuals unable to exercise entirely, e.g., lower extremity amputations without feasible alternatives for adapted exercise
6. Having severe musculoskeletal pain at rest or with minimal activity
7. Unable to sit, stand or walk unassisted (walking device such as cane or walker allowed)
8. Having shortness of breath at rest or with activities of daily living (NYHAClass IV)
9. Individuals with exercise participation ≥ 3 times per week that addressed ≥ 2 of the domains
10. Myocardial infarction within the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 Month
  Determining recruitment by eligible number/enrolled number
Retention rate | 3 Months
  Determining retention rate by patients who completed visit 2 / recruited patients
Adherence rate | 3 Months
  Determining the adherence by the number of participation in exercise sessions by a participant / the number of the exercise sessions planned in the program
Goal Achievement Scale (GAS) | Pre-test and 3 Months Later (Post-test)
  Using GAS to individually evaluate the effect of the intervention, accounting for differences in disease stages and personalized goals.

SECONDARY OUTCOMES:
Rate of changes of daily physical activity level | Pre-test and 3 Months Later (Post-test)
  To examine the effect of home-based synchronous tele-exercise on daily activity level by using Low Physical activity questionnaire.
  The questionnaire consists of 11 items that assess various parameters of physical activity within the past 7 days. These parameters include the amount of time spent walking around the neighborhood, for fitness or pleasure, and for transportation purposes, as well as the average duration of sedentary and sitting activities. The questionnaire also calculates the kilocalories expended during light, moderate, vigorous, and total physical activities.
Rate of changes of Frailty level | Pre-test and 3 Months Later (Post-test)
  To examine the effect of home-based synchronous tele-exercise on daily activity level by using Fried Frailty Index.
  Patients will be considered frail if they met 3 or more of the following 5 criteria: unintentional weight loss of 10 pounds or more in the prior year by self-report; exhaustion based on responses to two questions about energy; low physical activity based on the Minnesota questionnaire (< 383 kcal/wk for men or < 270 kcal/wk for women); slow gait speed (based on gender- and height-stratified cutoffs); and weak grip strength (based on gender- and BMI-stratified cutoffs). Patients will be asked whether they are independent in the following activities of daily living (ADLs): bathing, dressing, getting in and out of a chair, and walking around their home or apartment. Those reporting dependency in one or more will be considered to have an ADL limitation.
Rate of changes of physical function level | Pre-test and 3 Months Later (Post-test)
  To examine the effect of home-based synchronous tele-exercise on physical function level by 6 minute walk test and short physical performance battery test

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tabibi, Dr, Principal Investigator — Pardis Specialized Wellness Institute; Paul Bennett, Prof, Study Director — Griffith University; Farzad Nazemi, Study Director — Pardis Specialized Wellness Institute
Locations (1):
- Khorshid Dialysis Center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results reported in the published article will be shared after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date
Access Criteria: Not applicable. It will be accessible for public.

REFERENCES:
- [Background] Johansen KL, Kaysen GA, Dalrymple LS, Grimes BA, Glidden DV, Anand S, Chertow GM. Association of physical activity with survival among ambulatory patients on dialysis: the Comprehensive Dialysis Study. Clin J Am Soc Nephrol. 2013 Feb;8(2):248-53. doi: 10.2215/CJN.08560812. Epub 2012 Nov 2. PMID 23124787
- [Background] Delgado C, Johansen KL. Barriers to exercise participation among dialysis patients. Nephrol Dial Transplant. 2012 Mar;27(3):1152-7. doi: 10.1093/ndt/gfr404. Epub 2011 Jul 26. PMID 21795245
- [Background] Tao X, Chow SK, Wong FK. A nurse-led case management program on home exercise training for hemodialysis patients: A randomized controlled trial. Int J Nurs Stud. 2015 Jun;52(6):1029-41. doi: 10.1016/j.ijnurstu.2015.03.013. Epub 2015 Mar 26. PMID 25840898
- [Background] Painter PL, Nelson-Worel JN, Hill MM, Thornbery DR, Shelp WR, Harrington AR, Weinstein AB. Effects of exercise training during hemodialysis. Nephron. 1986;43(2):87-92. doi: 10.1159/000183805. PMID 3713951
- [Background] Barcellos FC, Santos IS, Umpierre D, Bohlke M, Hallal PC. Effects of exercise in the whole spectrum of chronic kidney disease: a systematic review. Clin Kidney J. 2015 Dec;8(6):753-65. doi: 10.1093/ckj/sfv099. Epub 2015 Oct 20. PMID 26613036
- [Background] Baggetta R, D'Arrigo G, Torino C, ElHafeez SA, Manfredini F, Mallamaci F, Zoccali C, Tripepi G; EXCITE Working group. Effect of a home based, low intensity, physical exercise program in older adults dialysis patients: a secondary analysis of the EXCITE trial. BMC Geriatr. 2018 Oct 20;18(1):248. doi: 10.1186/s12877-018-0938-5. PMID 30342464
- [Background] Hiraki K, Shibagaki Y, Izawa KP, Hotta C, Wakamiya A, Sakurada T, Yasuda T, Kimura K. Effects of home-based exercise on pre-dialysis chronic kidney disease patients: a randomized pilot and feasibility trial. BMC Nephrol. 2017 Jun 17;18(1):198. doi: 10.1186/s12882-017-0613-7. PMID 28623895
- [Background] Darawad MW, Khalil AA. Jordanian dialysis patients' perceived exercise benefits and barriers: a correlation study. Rehabil Nurs. 2013 Nov-Dec;38(6):315-22. doi: 10.1002/rnj.98. Epub 2013 May 23. PMID 23703743
- [Background] Rosa CS, Bueno DR, Souza GD, Gobbo LA, Freitas IF Jr, Sakkas GK, Monteiro HL. Factors associated with leisure-time physical activity among patients undergoing hemodialysis. BMC Nephrol. 2015 Nov 27;16:192. doi: 10.1186/s12882-015-0183-5. PMID 26613791
- [Background] Bennett PN, Bohm C, Harasemiw O, Brown L, Gabrys I, Jegatheesan D, Johnson DW, Lambert K, Lightfoot CJ, MacRae J, Meade A, Parker K, Scholes-Robertson N, Stewart K, Tarca B, Verdin N, Wang AY, Warren M, West M, Zimmerman D, Li PK, Thompson S. Physical activity and exercise in peritoneal dialysis: International Society for Peritoneal Dialysis and the Global Renal Exercise Network practice recommendations. Perit Dial Int. 2022 Jan;42(1):8-24. doi: 10.1177/08968608211055290. Epub 2021 Nov 7. PMID 34743628
- [Background] Myers J, Chan K, Chen Y, Lit Y, Patti A, Massaband P, Kiratli BJ, Tamura M, Chertow GM, Rabkin R. Effect of a Home-Based Exercise Program on Indices of Physical Function and Quality of Life in Elderly Maintenance Hemodialysis Patients. Kidney Blood Press Res. 2021;46(2):196-206. doi: 10.1159/000514269. Epub 2021 Mar 26. PMID 33774634
- [Background] Ortega-Perez de Villar L, Martinez-Olmos FJ, Perez-Dominguez FB, Benavent-Caballer V, Montanez-Aguilera FJ, Mercer T, Segura-Orti E. Comparison of intradialytic versus home-based exercise programs on physical functioning, physical activity level, adherence, and health-related quality of life: pilot study. Sci Rep. 2020 May 19;10(1):8302. doi: 10.1038/s41598-020-64372-y. PMID 32427935
- [Background] Manfredini F, Mallamaci F, D'Arrigo G, Baggetta R, Bolignano D, Torino C, Lamberti N, Bertoli S, Ciurlino D, Rocca-Rey L, Barilla A, Battaglia Y, Rapana RM, Zuccala A, Bonanno G, Fatuzzo P, Rapisarda F, Rastelli S, Fabrizi F, Messa P, De Paola L, Lombardi L, Cupisti A, Fuiano G, Lucisano G, Summaria C, Felisatti M, Pozzato E, Malagoni AM, Castellino P, Aucella F, Abd ElHafeez S, Provenzano PF, Tripepi G, Catizone L, Zoccali C. Exercise in Patients on Dialysis: A Multicenter, Randomized Clinical Trial. J Am Soc Nephrol. 2017 Apr;28(4):1259-1268. doi: 10.1681/ASN.2016030378. Epub 2016 Dec 1. PMID 27909047
- [Background] Velayati F, Ayatollahi H, Hemmat M. A Systematic Review of the Effectiveness of Telerehabilitation Interventions for Therapeutic Purposes in the Elderly. Methods Inf Med. 2020 May;59(2-03):104-109. doi: 10.1055/s-0040-1713398. Epub 2020 Jul 6. PMID 32629502
- [Background] Laver KE, Schoene D, Crotty M, George S, Lannin NA, Sherrington C. Telerehabilitation services for stroke. Cochrane Database Syst Rev. 2013 Dec 16;2013(12):CD010255. doi: 10.1002/14651858.CD010255.pub2. PMID 24338496
- [Background] Zhao Y, Chung PK, Tong TK. Effectiveness of a balance-focused exercise program for enhancing functional fitness of older adults at risk of falling: A randomised controlled trial. Geriatr Nurs. 2017 Nov-Dec;38(6):491-497. doi: 10.1016/j.gerinurse.2017.02.011. Epub 2017 Mar 27. PMID 28359614
- [Background] Marthick M, Dhillon HM, Alison JA, Cheema BS, Shaw T. An Interactive Web Portal for Tracking Oncology Patient Physical Activity and Symptoms: Prospective Cohort Study. JMIR Cancer. 2018 Dec 21;4(2):e11978. doi: 10.2196/11978. PMID 30578217
- [Background] Marthick M, McGregor D, Alison J, Cheema B, Dhillon H, Shaw T. Supportive Care Interventions for People With Cancer Assisted by Digital Technology: Systematic Review. J Med Internet Res. 2021 Oct 29;23(10):e24722. doi: 10.2196/24722. PMID 34714246
- [Background] Marthick M, Janssen A, Cheema BS, Alison J, Shaw T, Dhillon H. Feasibility of an Interactive Patient Portal for Monitoring Physical Activity, Remote Symptom Reporting, and Patient Education in Oncology: Qualitative Study. JMIR Cancer. 2019 Nov 28;5(2):e15539. doi: 10.2196/15539. PMID 31778123
- [Background] Rifkin DE, Abdelmalek JA, Miracle CM, Low C, Barsotti R, Rios P, Stepnowsky C, Agha Z. Linking clinic and home: a randomized, controlled clinical effectiveness trial of real-time, wireless blood pressure monitoring for older patients with kidney disease and hypertension. Blood Press Monit. 2013 Feb;18(1):8-15. doi: 10.1097/MBP.0b013e32835d126c. PMID 23275313
- [Background] Ishani A, Christopher J, Palmer D, Otterness S, Clothier B, Nugent S, Nelson D, Rosenberg ME; Center for Innovative Kidney Care. Telehealth by an Interprofessional Team in Patients With CKD: A Randomized Controlled Trial. Am J Kidney Dis. 2016 Jul;68(1):41-9. doi: 10.1053/j.ajkd.2016.01.018. Epub 2016 Mar 2. PMID 26947216
- [Background] Reese PP, Bloom RD, Trofe-Clark J, Mussell A, Leidy D, Levsky S, Zhu J, Yang L, Wang W, Troxel A, Feldman HI, Volpp K. Automated Reminders and Physician Notification to Promote Immunosuppression Adherence Among Kidney Transplant Recipients: A Randomized Trial. Am J Kidney Dis. 2017 Mar;69(3):400-409. doi: 10.1053/j.ajkd.2016.10.017. Epub 2016 Dec 7. PMID 27940063
- [Background] McGillicuddy JW, Gregoski MJ, Weiland AK, Rock RA, Brunner-Jackson BM, Patel SK, Thomas BS, Taber DJ, Chavin KD, Baliga PK, Treiber FA. Mobile Health Medication Adherence and Blood Pressure Control in Renal Transplant Recipients: A Proof-of-Concept Randomized Controlled Trial. JMIR Res Protoc. 2013 Sep 4;2(2):e32. doi: 10.2196/resprot.2633. PMID 24004517